CLINICAL TRIAL: NCT07173829
Title: A Prospective Study to Better Understand the Molecular, Immune and Metabolic Mechanisms Involved in Glioblastoma Recurrence and Progression, in the Aim to Identify New Therapeutic Targets and to Improve Current Therapies
Brief Title: A Study to Better Understand the Biological and Molecular Mechanisms Involved in Glioblastoma Recurrence and Progression
Acronym: BORDEAUX-GLIO
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: University of Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/06
Record Dates: First submitted 2023-08-02; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma
Keywords: Glioblastoma progression; Glioblastoma recurrence; Metabolism; Lactate; Metabolomic; Transcriptomic; Radiation therapy; Radiosensitizer; Immunotherapy; γδ T lymphocytes
MeSH Terms: conditions — Glioblastoma | interventions — Sampling Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood Cerebral brain tumor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Recruited patient: Glioblastoma patient with indication for neurosurgery
  Interventions: Other: samples

INTERVENTIONS:
Other: samples — A 50 ml blood sample will be taken from the patient before the operation, and two 0.3 cm3 tumor samples will be taken during the operation from the resected tumor.

SUMMARY:
BORDEAUX-GLIO is a prospective, monocentric study which will describe the molecular, immune and metabolic pathways involved in the progression and relapse of glioblastoma, using blood and tumor samples from patients who have undergone surgery for newly diagnosed or recurrent glioblastoma in the center.

DETAILED DESCRIPTION:
Glioblastoma is the most common and aggressive primary brain tumor in adults, whose relapse is almost systematic despite surgery, radiation therapy and temozolomide (STUPP protocol). Several clinical trials evaluating targeted therapy and immune checkpoint inhibitors have led to disappointed results. There is an unmet need to better understand the molecular and immune mechanisms underlying the invasion and progression of these tumors, in order to identify new therapeutic targets. The Bordeaux University Hospital is a leading French treatment center for glioblastoma, providing a large number of biological samples that can be analyzed at the molecular, immune and metabolic levels by specialized local teams.

Tumor tissue will be collected during patient surgery from primitive or recurrent glioblastoma, as well as blood samples, to perform transcriptomic and metabolomic analysis, including spatial transcriptomic and metabolomic, ex vivo generation of γδT lymphocytes and patient-derived xenografts.

A secondary objective is to develop, in preclinical models, innovative drugs with radiosensitizing effect and a γδT cell immunotherapy active against glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 years or older, with highly suspected glioblastoma on neuro-imagery
* Planned surgical tumor resection,
* No objection to participate in research
* Signed genetic consent

Exclusion Criteria:

* Patients under guardianship, curatorship or protective supervision
* Taking immunosuppressants
* Pregnant or breast-feeding women
* Patients deprived of their liberty by judicial or administrative decision, or under psychiatric care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of 18 years or older, with highly suspected glioblastoma on neuro-imagery
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Molecular mechanism | at inclusion (T0)
  Description of the molecular mechanism involved in the progression and recurrence of glioblastoma
Metabolic mechanism | at inclusion (T0)
  Description of the metabolic mechanism involved in the progression and recurrence of glioblastoma.
Immune mechanism | at inclusion (T0)
  Description of the immune mechanism involved in the progression and recurrence of glioblastoma

CONTACTS AND LOCATIONS:
Overall Officials: Julien ENGELHARDT, Dr, Principal Investigator — University Hospital, Bordeaux; Mathieu LARROQUETTE, Dr, Study Chair — University Hospital, Bordeaux; Guillaume CHOTARD, Dr, Study Chair — University Hospital, Bordeaux; Lionel COUZI, Pr, Study Chair — Bordeaux university Hospital, Bordeaux University; Andreas BIKFALVI, Pr, Study Chair — University of Bordeaux; Charles DUPIN, Dr, Study Chair — University Hospital, Bordeaux; Véronique VENDRELY, Pr, Study Chair — Bordeaux university Hospital, Bordeaux University; Julie DECHANET-MERVILLE, Dr, Study Chair — University of Bordeaux; Thomas DAUBON, Dr, Study Chair — University of Bordeaux

IPD SHARING:
Plan to Share IPD: No